CLINICAL TRIAL: NCT01160263
Title: Study of Dopamine and Serotonin Transporters in Patients With Amyotrophic Lateral Sclerosis and Controls. Analysis With 123I-FP-CIT (Datscan) and 123I-ADAM Brain SPECT
Brief Title: Study of Dopamine and Serotonin Transporters in Patients With Amyotrophic Lateral Sclerosis and Controls
Acronym: DOSERAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); ARS (Association pour la Recherche sur la Sclérose Latérale Amyotrophique) (Unknown); Agence Générale des Equipements et Produits de Santé (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P080402; P080402 (Other: DRCD); AOM 07225 (Other: DRCD)
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; serotonin; dopamine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ioflupane; 2-((2-((dimethylamino)methyl)phenyl)thio)-5-iodophenylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- patients without stiffness (Other)
  Interventions: Drug: SPECT : 123 I-FP-CIT (DATSCAN) and 123I-ADAM
- patients with pyramidal stiffness (Other)
  Interventions: Drug: SPECT : 123 I-FP-CIT (DATSCAN) and 123I-ADAM
- patients with mixed stiffness (Other)
  Interventions: Drug: SPECT : 123 I-FP-CIT (DATSCAN) and 123I-ADAM

INTERVENTIONS:
Drug: SPECT : 123 I-FP-CIT (DATSCAN) and 123I-ADAM — 123 I-FP-CIT (DATSCAN) : 185 MBq (5 mCi), 2,5 ml will be injected via an arm intravenous catheter.
  123I-ADAM:185 MBq,5 ml will be injected via an arm intravenous catheter.
  Other Names: PECT : 123 I-FP-CIT (DATSCAN) and 123I-ADAM

SUMMARY:
The purpose of this study is to study the transporters of serotonin and dopamine in ALS patients in relation with the clinical phenotype, i.e., patients without stiffness, patients with pyramidal stiffness, patients with mixed (pyramidal and extra pyramidal) stiffness.

For such a goal the investigators will use SPECT to compare the binding of two specific tracers in ALS patients and in matched healthy controls.

DETAILED DESCRIPTION:
Study design This study is a prospective cross-sectional controlled multicentric clinical study in 60 ALS patients and 20 controls.

Three cohorts of 20 ALS patients(patients without stiffness, patients with pyramidal stiffness, patients with mixed pyramidal and extra pyramidal stiffness) and 20 healthy controls will be included in this study

Study centres 40 ALS patients and 13 controls will be included in the Paris ALS center, 20 ALS patients and 7 controls will be included in the Tours ALS center.

MRI will be performed at the Neuroradiology department of salpetriere hospital (Paris) and Bretonneau hospital (Tours) SPECT will be done in the nuclear medicine center of each hospital (Paris- Tours).

Study duration Per patient or control, the study will be lasted one month. The total study duration will be two years

ELIGIBILITY:
Inclusion Criteria:

1. Patients (men or women)

   * between 39 (exclusive) and 66 (inclusive) years old
   * with a sporadic ALS, defined, probable or laboratory possible
   * with a disease duration between 3 months (inclusive) and 5 years (exclusive)
   * treated with rilutek at 100 mg/ day since at least 1 month
2. Patients will be assigned in three groups in relation with the clinical phenotypes:

   * 20 patients without stiffness
   * 20 patients with pyramidal stiffness (spasticity patients).
   * 20 patients with mixed stiffness (both spasticity and rigidity).
3. Patients have to be capable of thoroughly understanding the information given; have signed the informed consent form (signature of spouse or family relative or acceptable third party is acceptable if the patient is physically unable to sign).
4. To have social insurance

Exclusion Criteria:

1. Patients with a FRONTO temporal dementia (according to NEARY' criteria)
2. Patients with any concomitant life-threatening disease or any disease or impairment likely to interfere with functional assessment;
3. Patients with any major evolving psychiatric disorder or major anxiety disorder according to DSM-IV criteria (APA, 1996)
4. Patients receiving treatments which could interfere with the serotonin or dopamine metabolism
5. Patients with contraindications for the dat-scan and /or ADAM scan
6. Patients with contraindications for the MRI scan.
7. Patients with previous vascular, traumatic or tumoral cerebral lesions making impossible the quantification of the tracer
8. Patients with a cancer within the past 5
9. Patients child bearing, breast feeding or in the second part of their cycle without any efficient contraceptive device or treatment
10. Patients liable not to be co-operative or comply with the trial requirements (as assessed by the investigator), or unable to be reached in the event of an emergency;

Ages: 39 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Dopamine transporter binding potential | 1 month

SECONDARY OUTCOMES:
Serotonin transporter binding potential | 1 month
Relationships between transporter binding potential and the clinical scores | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Lucette Lacomblez, MD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (2):
- France (2):
  - Salpêtrière Hospital, Paris
  - Bretonneau Hospital, Tours